CLINICAL TRIAL: NCT02354950
Title: A Phase I Study to Evaluate the Pharmacokinetics and Safety of GSK1265744 in Subjects With Hepatic Impairment and Healthy Matched Control Subjects
Brief Title: A Study to Evaluate Pharmacokinetic (PK) and Safety of GSK1265744 in Subjects With Hepatic Impairment and Control Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201479
Record Dates: First submitted 2015-01-29; First posted 2015-02-03 (Estimated); Last update posted 2020-08-05 (Actual); Status verified 2020-08

CONDITIONS: HIV Infections
Keywords: GSK1265744; healthy controls; pharmacokinetic; Hepatic Impairment
MeSH Terms: conditions — HIV Infections | interventions — cabotegravir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part 1 Cohort 1 (Moderate hepatic impairment subjects) (Experimental): Subjects with moderate hepatic impairment will receive GSK1265744 30mg as a single oral dose in the fasted state followed by pharmacokinetic sampling for total concentrations of GSK1265744 in plasma
  Interventions: Drug: GSK1265744 30mg
- Part 1 Cohort 2 (Healthy control subjects) (Experimental): Healthy control subjects will receive GSK1265744 30mg as a single oral dose in the fasted state followed by pharmacokinetic sampling for total concentrations of GSK1265744 in plasma
  Interventions: Drug: GSK1265744 30mg
- Part 2 Cohort 3 (Mild hepatic impairment subjects) (Experimental): Subjects with mild hepatic impairment will receive GSK1265744 30mg as a single oral dose in the fasted state followed by pharmacokinetic sampling for total concentrations of GSK1265744 in plasma
  Interventions: Drug: GSK1265744 30mg
- Part 2 Cohort 4 (Healthy control subjects) (Experimental): Healthy control subjects will receive GSK1265744 30mg as a single oral dose in the fasted state followed by pharmacokinetic sampling for total concentrations of GSK1265744 in plasma
  Interventions: Drug: GSK1265744 30mg

INTERVENTIONS:
Drug: GSK1265744 30mg — GSK1265744 30mg tablets are white to almost white coated oval tablets. All subjects will receive GSK1265744 30mg as a single oral dose in the fasted state followed by PK sampling.

SUMMARY:
This will be a Phase 1, open-label, parallel group, two-part, single-dose adaptive study in adults with moderate and mild (if needed) hepatic impairment and matched, healthy control subjects with normal hepatic function. In Part 1, healthy control subjects (n=8) matched to subjects with moderate (n=8) hepatic impairment will be enrolled. If the geometric mean total plasma area under the concentration-time curve from time zero (pre-dose) extrapolated to infinite time (AUC[0-infinity]) of GSK1265744 is increased by >2-fold in moderately impaired subjects relative to matched controls, Part 2 will be conducted to evaluate GSK1265744 PK in subjects with mild hepatic impairment (n=8) and matched, control subjects (n=8). All subjects will receive a single 30 milligram (mg) oral dose of GSK1265744. The primary objective of the study is to compare plasma PK parameters of GSK1265744 in subjects with hepatic impairment to healthy controls matched in gender, age, and body mass index (BMI).

ELIGIBILITY:
Inclusion Criteria:

* Hepatic Impaired Subjects (Cohort 1 and 3)
* Between 18 and 70 years of age

Part 1 subjects with Moderate Hepatic Impairment Only (Cohort 1):

* Subject is considered to have moderate hepatic impairment (of any etiology) and has been clinically stable for at least 1 month prior to screening. Having moderate hepatic impairment with a Child-Pugh score of 7-9 and previous confirmation of liver cirrhosis.

Part 2 subjects with Mild Hepatic Impairment Only (Cohort 3):

* Subject is considered to have mild hepatic impairment (of any etiology) and has been clinically stable for at least 1 month prior to screening. Having mild hepatic impairment, with a Child-Pugh score of 5-6 and previous confirmation of chronic liver disease.
* Supplemental inclusion criteria for all hepatically impaired subjects: Chronic (>6 months), stable (no acute episodes of illness within the previous 1 month prior to screening due to deterioration in hepatic function) hepatic impairment due to any etiology. Subjects must also remain stable throughout the Screening period. - Body weight >=50 kilogram (kg) and BMI within the range 19 - 41 kilogram per meter square (kg/m^2) (inclusive).
* Male or female: Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the consent form and the protocol.

Inclusion Criteria for Healthy Subjects (Cohorts 2 and 4):

* Healthy control subjects will be matched for age +/-10 years to subjects in the respective hepatic impairment cohort but must also remain in the age range between 18 and 70 years inclusive, at the time of signing the informed consent.
* Healthy as determined by the investigator or medically qualified designee. Healthy control subjects will be matched for BMI +/-25 percent to subjects in the respective hepatic impairment cohort but must also remain in the range of: Body weight >=50 kg and BMI within the range 19 - 41 kg/m^2 (inclusive)
* Male or female: Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the consent form and in the protocol.

Exclusion Criteria:

* Exclusion Criteria for Hepatic Impaired Subjects (Cohort 1 and 3):
* Presence of Grade 3 or 4 elevations in aspartate aminotransferase (AST), alanine aminotransferase (ALT), or bilirubin; corrected QT interval (QTc) > 480 milliseconds (msec);
* The subject's systolic BP is outside the range of 90-160 millimeter of mercury (mmHg), or diastolic BP is outside the range of 45-95mmHg or heart rate is outside the range of 50-100 beats per minute (bpm) for female subjects or 45-100 bpm for male subjects
* Evidence of previous myocardial infarction in the past 12 months or any clinically significant active cardiovascular disease that, in the opinion of the investigator, could interfere with the safety of the subject.
* Any clinically significant conduction abnormality
* Any significant arrhythmia.
* Non-sustained or sustained ventricular tachycardia.
* Evidence of recent infection with Hepatitis B and/or Hepatitis C within preceding 6 months. Subjects with chronic Hepatitis B or C (duration>6 months)
* Subjects with a pre-existing condition (except hepatic impairment) interfering with normal gastrointestinal anatomy or motility that could interfere with the absorption, metabolism, and/or excretion of the study drugs. Subjects with a history of cholecystectomy and inflammatory bowel disease should be excluded.

Subjects with a history of peptic ulceration or pancreatitis within the preceding 6 months of screening should be excluded.

* Subjects with previous gastrointestinal (GI) surgery (except appendectomy more than three months prior to study) should be excluded.
* Subjects with creatinine clearance (CLCR) <=60 milliliter per minute (mL/min) (calculated by the Modification of Diet in Renal Disease [MDRD] equation).
* Subjects with advanced ascites (Grade 3 or 4).
* Subjects with refractory encephalopathy as judged by the investigator or significant Central Nervous System (CNS) disease.
* History of gastric or esophageal variceal bleeding within the past 6 months;
* Subjects with Transjugular Intrahepatic Portosystemic Shunt (TIPS) placement;
* Presence of hepatopulmonary or hepatorenal syndrome;
* Presence of primarily cholestatic liver diseases;
* History of liver transplantation;
* Subjects with signs of active infection;
* Subjects with unstable cardiac function or subjects with hypertension whose blood pressure is not controlled;
* Diabetic subjects whose diabetes is not controlled;
* Subjects with any other medical condition (other than hepatic impairment) which, in the judgment of the investigator and medical monitor, could jeopardize the integrity of the data derived from that subject or the safety of the subject;
* Subjects requiring any concurrent prohibited medication listed in study protocol;
* Subjects receiving lactulose who are medically unable to halt lactulose administration from 8 hours before dosing with study drug to 4 hours after dosing with study drug;
* Subjects with a change in dose regimen of medically required medication within the 2 weeks prior to dosing;
* History of regular alcohol consumption within 6 months of the study;
* Inability or unwillingness to comply with lifestyle and/or dietary restrictions outlined in protocol;
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or Medical Monitor, contraindicates their participation. ;
* Unwillingness or inability to follow the procedures outlined in the protocol;
* A positive pre-study drug/alcohol screen;
* A positive test for human immunodeficiency virus (HIV) antibody;
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period;
* Subject's with a platelet count <50,000 x 10^9 per liter (/L) of blood who have had a major bleeding episode within the past 6 months;
* Subjects with electrolyte imbalance;
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exclusion Criteria for Healthy Subjects (Cohorts 2 and 4):
* ALT and bilirubin >1.5x upper limit of normal (ULN) (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35 percent). A single repeat is allowed for eligibility determination;
* Current or chronic history of liver disease;
* QTc > 450 msec;
* Exclusion criteria for screening ECG as per study protocol;
* Systolic BP outside the range of 90-145 mmHg, or diastolic BP outside the range of 45-95 mmHg or heart rate outside the range of 50-100 bpm for female subjects or 45-100 bpm for male subjects;
* Evidence of previous myocardial infarction;
* Any clinically significant conduction abnormality;
* Any significant arrhythmia.
* Non-sustained or sustained ventricular tachycardia;
* Subjects with a pre-existing condition interfering with normal gastrointestinal anatomy or motility that could interfere with the absorption, metabolism, and/or excretion of the study drugs. Subjects with a history of cholecystectomy and inflammatory bowel disease. Subjects with a history of peptic ulceration or pancreatitis within 6 months of screening. Subjects with previous GI surgery (except appendectomy more than three months prior to study).
* The use of any concurrent prohibited medications as outlined in study protocol.
* History of regular alcohol consumption within 6 months of the study,
* Inability or unwillingness to comply with lifestyle and/or dietary restrictions outlined in study protocol.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or Medical Monitor, contraindicates their participation.
* Unwillingness or inability to follow the procedures outlined in study protocol.
* Presence of hepatitis B surface antigen (HBsAg) (or positive hepatitis B core antibody with negative hepatitis B surface antibody) or positive hepatitis C antibody test result.
* A positive pre-study drug/alcohol screen.
* A positive test for HIV antibody.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within 56 days.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2015-06-22 (Actual); Primary Completion 2016-09-16 (Actual); Study Completion 2016-09-16 (Actual)

PRIMARY OUTCOMES:
Plasma area under the concentration-time curve from time zero (pre-dose) extrapolated to infinite time [AUC(0-infinity)] following a single oral dose of GSK1265744 | Pre-dose (within 15 minutes prior to dose), 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 120, 168 hours post dose (Day 8)
  Plasma PK samples (2 mL of blood per sample) will be collected to measure GSK1265744 at the following time points: pre-dose (within 15 minutes prior to dose), 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 120, 168 hours post dose
Maximum observed concentration (Cmax) following a single oral dose of GSK1265744 | Pre-dose (within 15 minutes prior to dose), 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 120, 168 hours post dose (Day 8)
  Plasma PK samples (2 mL of blood per sample) will be collected to measure GSK1265744 at the following time points: pre-dose (within 15 minutes prior to dose), 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 120, 168 hours post dose

SECONDARY OUTCOMES:
Unbound concentration and unbound fraction in plasma of GSK1265744 at 2 and 24 hours post dose | Up to 24 hours post dose (Day 2)
  Blood samples will be collected to measure bound and unbound plasma GSK1265744 concentrations at 2 and 24 hours post dose
Composite of PK parameters including AUC(0-t), %AUCex, C24, t1/2, CL/F, tlag, tmax, and Vz/F following a single oral dose of GSK1265744 | Pre-dose (within 15 minutes prior to dose), 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 120, 168 hours post dose (Day 8)
  PK parameters including plasma area under the concentration-time curve from time zero (pre-dose) to last time of quantifiable concentration [AUC(0-t)], percentage of AUC(0-infinity) obtained by extrapolation (%AUCex), concentration observed at 24-hours post dose (C24), apparent terminal phase half-life (t1/2), apparent clearance (CL/F), lag time before observation of drug concentrations (tlag), time of occurrence of Cmax (tmax) and apparent terminal phase volume of distribution (Vz/F) following a single oral dose of GSK1265744
Adverse events (AEs) assessment | Up to Day 14
  An AE is any untoward medical occurrence in a subject or clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product
Composite of Clinical laboratory parameters including hematology, and clinical chemistry | Up to Day 14
  Assessment of Laboratory parameters will include hematology, and clinical chemistry
Electrocardiogram (ECG) monitoring | Up to Day 2
  12-lead ECGs will be performed with the subject in a semi-supine position having rested in this position for at least 10 minutes beforehand
Composite of Vital signs assessments will include measurement of temperature, systolic and diastolic blood pressure, heart rate and respiratory rate | Up to Day 14
  Vital signs will be measured in semi-supine position after 10 minutes rest and will include temperature, systolic and diastolic blood pressure (BP), heart rate (HR) and respiratory rate

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (3):
- United States (3):
  - GSK Investigational Site, Lakewood, Colorado
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Minneapolis, Minnesota

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com/Posting.aspx?ID=20361

REFERENCES:
- [Background] Shaik JSB, Ford SL, Lou Y, Zhang Z, Bakshi KK, Tenorio AR, Trezza C, Spreen WR, Patel P. A Phase 1 Study to Evaluate the Pharmacokinetics and Safety of Cabotegravir in Patients With Hepatic Impairment and Healthy Matched Controls. Clin Pharmacol Drug Dev. 2019 Jul;8(5):664-673. doi: 10.1002/cpdd.655. Epub 2019 Feb 27. PMID 30811880